CLINICAL TRIAL: NCT04765579
Title: Effects of Ultrasonography-guided 4in1 Block Application on Postoperative Analgesia in Patients Undergoing Knee Surgery
Brief Title: Investigation of the Effect of 4 in 1 Block Application on Postoperative Analgesia in Knee Surgeries.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyran Köksal, resident, Derince Training and Research Hospital
Other Study IDs: Seyran-Tez
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Visual Analogy Scala

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4in1: 4in1 block will be applied in the operation room
  Interventions: Behavioral: visual analogy scala
- medical: medical analgesics will be applied in the service
  Interventions: Behavioral: visual analogy scala

INTERVENTIONS:
Behavioral: visual analogy scala — We will investigate the effect of 4in1 block by questioning the vas score of the patients, its effect on quadriceps strength, and additional analgesia needs for 24 hours.

SUMMARY:
to investigate the effects of ultrasonography-guided 4in1 block application on postoperative analgesia in patients undergoing knee surgery. After knee surgeries performed with spinal anesthesia, 4in1 block will be applied in one group and medical analgesics will be applied in the service in the other group.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 18-60 ages
* who were informed about the study and accepted,
* who underwent knee surgery

Exclusion Criteria:

* ASA III-IV
* who are under general anesthesia
* who do not agree to participate in the study
* who are urgently operated

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: knee surgeries performed with spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
visuel analogue scale | 6 months
  0:No pain, 10:Very severe pain

IPD SHARING:
Plan to Share IPD: No